CLINICAL TRIAL: NCT01530529
Title: A Phase 1, Cross-Over, Single-Dose, Open-Label Study to Estimate the Relative Bioavailability of a Modified-Release Formulation of PF-05180999 Under Fed and Fasted Conditions in Healthy Adult Subjects
Brief Title: A Study to Assess the Relative Bioavailability of a Modified-Release Formulation of PF-05180999
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3441007; B3441007
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: PF-05180999; safety; pharmacokinetics; relative bioavailability; Mental Disorders; Schizophrenia and Disorders with Psychotic Features; Schizophrenia
MeSH Terms: conditions — Mental Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-05180999 Immediate-Release (Experimental)
  Interventions: Drug: PF-05180999
- PF-05180999 Modified-Release 1 (Experimental)
  Interventions: Drug: PF-05180999
- PF-05180999 Modified-Release 2 (Experimental)
  Interventions: Drug: PF-05180999
- PF-05180999 Modified-Release 1 With Food (Experimental)
  Interventions: Drug: PF-05180999

INTERVENTIONS:
Drug: PF-05180999 — Single dose of 30 mg of PF-05180999 administered to fasted subjects as an immediate-release powder-in-capsule formulation
  Arms: PF-05180999 Immediate-Release
Drug: PF-05180999 — Single dose of 30 mg of PF-05180999 administered to fasted subjects as a modified-release formulation
  Arms: PF-05180999 Modified-Release 1
Drug: PF-05180999 — Single dose of 120 mg of PF-05180999 administered to fasted subjects as a modified-release formulation
  Arms: PF-05180999 Modified-Release 2
Drug: PF-05180999 — Single dose of 30 mg of PF-05180999 administered to fed subjects as a modified-release formulation
  Arms: PF-05180999 Modified-Release 1 With Food

SUMMARY:
The purpose of this study is to assess the bioavailability, safety, and tolerability of a modified-release formulation of PF-05180999 relative to an immediate-release formulation in healthy adult subjects. Two doses of the modified-release formulation and one dose of the immediate-release formulation will be evaluated under fasted conditions. One dose of the modified-release formulation will also be evaluated in the presence of food.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential

Exclusion Criteria:

* Evidence of clinically-significant medical illness, history of seizures, any condition possibly affecting drug absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of each Period
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of each Period
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of each Period
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of each Period
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post-dose of each Period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3441007&StudyName=A%20Study%20to%20Assess%20the%20Relative%20Bioavailability%20of%20a%20Modified-Release%20Formulation%20of%20PF-05180999